CLINICAL TRIAL: NCT01257022
Title: Preventing Drug Abuse and HIV in Hispanic First Offenders
Brief Title: Familias Unidas: Preventing Drug Abuse and HIV in Hispanic First Offenders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA025894-01 (NIH)
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Substance Use; Unsafe Sexual Behavior
Keywords: Prevention; HIV; Substance use; Hispanic; Adolescents; Unsafe sexual behavior; Behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Function Intervention (Experimental): Familias Unidas Intervention Program
  Interventions: Behavioral: Familias Unidas
- Treatment as Usual (No Intervention): Control

INTERVENTIONS:
Behavioral: Familias Unidas — There will be 8 group sessions and 4 family visits. During the group sessions, the facilitator offers support for parents and gently corrects maladaptive interactions between parents and adolescents. During family visits, facilitators assist families in practicing skills and restructuring family interactions. The parent group sessions focus on parental investment in the adolescent's worlds (e.g., peer and school worlds), family communication, family support, behavior management/positive parenting, parental monitoring, adolescent substance use, and adolescent unsafe sex and HIV.
  Arms: Family Function Intervention

SUMMARY:
The main goal of the proposed study is to evaluate the efficacy of Familias Unidas (United Families), a family-based, ecodevelopmental intervention found to be previously efficacious in preventing and reducing behavior problems, illicit drug use, and unsafe sexual behavior in non-delinquent Hispanic adolescents (Pantin et al., 2003; Prado, Pantin, Briones et al., 2007).

The study hypotheses are as follows:

Hypothesis 1. Familias Unidas will be more efficacious than Treatment as Usual in preventing drug use among Hispanic first offending adolescents or those who are at risk for committing a first time offense over time.

Hypothesis 1a. The effect of Familias Unidas on drug use will be partially mediated by improvements in family functioning.

Hypothesis 2. Familias Unidas will be more efficacious than Treatment as Usual in preventing unsafe sexual behavior among Hispanic first offending adolescents or those who are at risk for committing a first time offense over time.

Hypothesis 2a. The effect of Familias Unidas on unsafe sexual behavior will be partially mediated by improvements in family functioning.

Hypothesis 3. Familias Unidas will be more efficacious than Treatment as Usual in preventing subsequent criminal offenses among Hispanic first offending adolescents or in preventing a first time offense for those at risk for committing a first time offense over time.

Hypothesis 3a. The effect of Familias Unidas on subsequent criminal offenses will be mediated by family functioning.

DETAILED DESCRIPTION:
Familias Unidas aims to prevent drug use and unprotected sexual behavior by increasing family functioning. A sample of 240 Hispanic adolescent first offenders or those at risk of becoming first offenders (age range 12 to 17) and 240 primary caregivers will be randomized to one of two conditions: Familias Unidas or Treatment as Usual. The investigators do not expect any risks to participants for participating in this study; however, participants may feel embarrassed by some of the content or feel fatigued as a result of completing the assessments. Also, depending on which group participants are assigned to, they may be less likely to use drugs and practice unsafe sexual behaviors and more likely to function better as families.

The proposed study will be guided by four aims. AIM 1 is to evaluate the efficacy of Familias Unidas, relative to Treatment as Usual in preventing illicit drug use in a sample of Hispanic youth first offenders or those at high risk of committing a first offense; AIM 2 is to evaluate the efficacy of Familias Unidas, relative to Treatment as Usual in preventing unsafe sexual behavior; AIM 3 is to evaluate the efficacy of Familias Unidas, relative to Treatment as Usual in preventing a first offense or reducing the number of subsequent criminal offenses ; and AIM 4 is to assess the extent to which family functioning mediates the effects of the intervention on illicit drug use, unsafe sexual behavior, and first or subsequent criminal offenses.

Compared to non-Hispanic whites, Hispanic adolescents are highly vulnerable to drug use and HIV infection. Hispanic adolescents between the ages of 13 to 19 are five times more likely to be infected with HIV than are same-aged non-Hispanic Whites (CDC-P, 2006). Compared to non-Hispanic whites and to African Americans, Hispanic 8th graders report the highest lifetime, annual, and 30-day prevalence rates of alcohol, cigarette, and licit or illicit drug use (with the exception of amphetamines; Johnston et al., 2008). Hispanic adolescents also have higher rates of unprotected sex at last intercourse (CDC-P, 2007) than non-Hispanic whites or African Americans. Drug use and unsafe sexual behavior are risks for HIV infection. Hispanics are also a youthful population, with more than one-third under the age of 18 (Marotta & Garcia, 2003). Preventing drug use and HIV in Hispanics, and particularly among Hispanic youth at elevated risk for drug use and unsafe sexual behavior, such as Hispanics in the criminal justice setting or those at risk of entering the criminal justice system (Telpin, 2003), is therefore of vital importance.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male adolescents of Hispanic immigrant origin, defined by at least one parent born in a Spanish-speaking country of the Americas
2. First-time offenders or Hispanic adolescents, identified by Miami Dade County Public Schools as exhibiting Level III behaviors which include: assault/threat against a non-staff member, breaking and entering/burglary, fighting (serious), hazing, possession or use of alcohol and/or controlled substances, possession of simulated weapons, trespassing, and vandalism.
3. Adolescents between 12 and 17 years of age
4. Adolescents living with an adult primary caregiver who is willing to participate

Exclusion Criteria:

(a) Family reports to have (tentative or firm) plans to move out of the South Florida area during the year of the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Substance use | 1 year
  Substance use as measured by items similar to those in the Monitoring the Future Survey.
Unsafe sexual behavior | 1 year
  Unsafe sexual beahvior including unprotected sexual behavior and having sex while under the influence of alcohol or drugs.

SECONDARY OUTCOMES:
Family functioning | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Center for Family Studies and Miami-Dade County, Miami, Florida, United States

REFERENCES:
- [Derived] Prado G, Pantin H, Huang S, Cordova D, Tapia MI, Velazquez MR, Calfee M, Malcolm S, Arzon M, Villamar J, Jimenez GL, Cano N, Brown CH, Estrada Y. Effects of a family intervention in reducing HIV risk behaviors among high-risk Hispanic adolescents: a randomized controlled trial. Arch Pediatr Adolesc Med. 2012 Feb;166(2):127-33. doi: 10.1001/archpediatrics.2011.189. Epub 2011 Oct 3. PMID 21969363